CLINICAL TRIAL: NCT07109791
Title: Developing a National Approach to Surveillance and Prevention for Neonatal Ventilator-Associated Pneumonia
Brief Title: National Surveillance and Prevention of Neonatal VAP
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other); University of British Columbia (Other); University of Toronto (Other); McGill University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00149177; 202409-197813 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ventilator-Associated Pneumonia (VAP), Neonatal; Bronchopulmonary Dysplasia (BPD); Antibiotic-Resistant Organisms (AROs); Health-Care Associated Infection (HAI)
Keywords: Preterm; Neonate; Neonatal intensive care unit (NICU); Ventilator-Associated Pneumonia (VAP); Healthcare-associated infections (HAI); Invasive mechanical ventilation (IMV); Bronchopulmonary dysplasia (BPD); Antibiotic-resistant organisms (AROs); Antimicrobial stewardship; Implementation science; Quality improvement (QI); Infection surveillance
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Bronchopulmonary Dysplasia; Cross Infection; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VLBW infants with VAP Diagnosis: The study population will include all VLBW infants (birth weight <1500g) admitted to participating tertiary NICUs in Canada with diagnoses of VAP at physicians' discretion.

SUMMARY:
The goal of this observational study is to improve how hospital-acquired lung infections (called ventilator-associated pneumonia, or VAP) are diagnosed, treated and prevented in very low birth weight (VLBW) infants, babies born very early (preterm) or very small who often require respiratory support in hospital's neonatal intensive care units (NICUs).

The main questions it aims to answer are:

* How often do very-low-birth-weight (VLBW) infants get ventilator-associated pneumonia (VAP) in hospitals across Canada?
* How often are these VAP infections caused by germs that are resistant to antimicrobials (also known as antimicrobial-resistant organisms or AROs)?
* What types of antimicrobial-resistant germs (AROs) are causing them?
* How are these infections being treated with antibiotics, and can we reduce unnecessary antibiotic use?
* Which diagnostic definition is the best and most accurate for diagnosing VAP in newborns, based on real patient data and expert agreement?
* Can we use this information to create clear, evidence-based guidelines that help hospitals prevent and treat VAP in the same, effective way?

Researchers will compare how different hospitals define, report, and manage VAP to devise a shared, evidence-based approach that will lead to more accurate diagnoses and better treatment and outcomes for neonatal VAP.

Researchers will:

* Use data already collected in hospital records (per existing standard of clinical care).
* Analyse how often VAP occurs, how it is diagnosed, and how it is treated
* Work with experts and hospitals to develop and implement a standard, evidence-based plan for diagnosing, managing and preventing VAP in newborns

The overarching goal is to create a clear, nationwide approach to ensure hospitals across Canada care for preterm babies in a standardized manner, reduce infection rates, avoid unnecessary antibiotic use, and improve outcomes for these vulnerable infants.

DETAILED DESCRIPTION:
PURPOSE: The purpose of this study is to develop neonatal-specific diagnostic criteria and management guidelines for VAP in VLBW infants in Canadian NICUs, and to improve clinical outcomes through better surveillance, diagnosis, management and antimicrobial stewardship.

HYPOTHESIS:

* We expect substantial variability in VAP incidence across the participating NICUs.
* We expect notable differences in the proportion of VAP events attributable to AROs and in the duration of antimicrobial treatment administered.

AIMS/OBJECTIVES:

1. Aim 1: To characterise neonatal VAP incidence by collecting data on infants diagnosed with VAP using three commonly applied definitions, while also identifying AROs, and evaluating patterns of antimicrobial use for VAP treatment across tertiary NICUs.
2. Aim 2: To identify the most appropriate, neonatal-specific VAP diagnostic definition by integrating systematically collected clinical data, statistical analyses, and expert consensus through Delphi methodology.
3. Aim 3: To translate these findings into practice by developing evidence-based clinical guidelines and tailored implementation strategies for VAP prevention and management.

STUDY POPULATION AND SAMPLE SIZE: The study population will include all VLBW infants (i.e., the group of infants neonates with the highest risk of infections within NICUs) admitted to participating tertiary NICUs in Canada with diagnoses of VAP at physicians' discretion.

RESEARCH METHODS: This project is a multi-centre prospective cohort study, conducted in collaboration with a network of tertiary NICUs in Canada.

ELIGIBILITY:
INCLUSION CRITERIA:

* All VLBW infants admitted to participating tertiary NICUs in Canada
* All neonatal VAP events diagnosed based on the physicians' discretion

EXCLUSION CRITERIA:

* Infants with major congenital anomalies
* Infants with moribund status on admission

Max Age: 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: STUDY POPULATION:
  The study population will include all VLBW infants admitted to participating tertiary NICUs in Canada from 2025-2028 inclusive, diagnosed with VAP at physicians' discretion during their admission.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
VAP Incidence | 2025-2028
  The number of VAP events per 1000 ventilator-days, per the three distinct definitions (Years 1-4).
  Unit of Measure: Number of VAP events

SECONDARY OUTCOMES:
Prevalence of VAP Among VLBW Infants | 2025-2028
  The proportion of VLBW infants with at least 1 episode of VAP Unit of Measure: Percentage of participants (%)
Other Adverse Outcomes | 2025-2028
  VAP Recurrence Rate Description: Proportion of participants who experience a recurrence of ventilator-associated pneumonia (VAP) during the study period Unit of Measure: Percentage of participants (%)
  Mortality Rate Description: Number of participants who die during the study period Unit of Measure: Number of participants
  Number of Participants Diagnosed with Bronchopulmonary Dysplasia (BPD) Description: Number of participants who develop BPD Unit of Measure: Number of participants
  Need for Invasive Mechanical Ventilation (IMV) at 36 Weeks Corrected Gestational Age Description: Number of participant
VAP Incidence Attributable to AROs | 2025-2028
  ARO-related VAP events; and the duration of antimicrobial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joseph Ting, Staff Neonatologist and Clinical Research Professor, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
due to data privacy and regulations

REFERENCES:
- [Derived] Li CZ, Tse-Chang A, Yoon EW, Paquette V, Roberts A, Afifi J, Yang CL, Khurshid F, Augustine S, Choudhury J, Elsharkawy A, Hamilton C, Hicks M, Joynt C, Wang D, Lee KS, Louis D, Robinson JL, Mohamed A, Mitra S, Shah VS, Srigley JA, Stavel M, Sherlock R, Wong J, Kuan MT, Madise-Wobo AD, Lemyre B, Joly C, Kharrat A, Gupta-Bhatnagar S, Zarembo M, Bacchini F, Beltempo M, Shah PS, Ting JY. Protocol for developing a national approach to surveillance and prevention for neonatal ventilator-associated pneumonia. BMJ Paediatr Open. 2026 Jan 12;10(1):e004234. doi: 10.1136/bmjpo-2025-004234. PMID 41526087